CLINICAL TRIAL: NCT02115477
Title: Prevalence, Complications and Risk Factors for Lymphedema After Pelvic and Paraaortic Lymphadenectomy in Primary Radical Surgery for Early Stage Endometrial Carcinoma.
Brief Title: Lymphedema After Primary Surgery for Endometrial Cancer
Acronym: LASEC
Status: Completed | Type: Observational
Sponsor: Preben Kjolhede, MD, professor (Other)
Collaborators: Swedish Cancer Society (Other); Medical Research Council of Southeast Sweden (Other Government); Ostergotland County Council, Sweden (Other); Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Preben Kjolhede, MD, professor, Professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Other Study IDs: Version 2013-09-22/2014-03-21; The Swedish Cancer Society (Other Grant/Funding Number: CAN 2013/620)
Record Dates: First submitted 2014-04-13; First posted 2014-04-16 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Carcinoma of the Endometrium; Hysterectomy; Lymphadenectomy
Keywords: Uterus cancer; Hysterectomy; Lymphadenectomy; Lymphedema
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Lymphedema | interventions — Lymph Node Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group with lymphadenectomy: The group of women with high risk endometrial cancer who undergoes pelvic and/or paraaortic lymphadenectomy at primary surgery
  Interventions: Procedure: Lymphadenectomy
- Group without lymphadenectomy: The group of women with low risk endometrial cancer who do not have lymphadenectomy at primary surgery

INTERVENTIONS:
Procedure: Lymphadenectomy — Pelvic and/or paraaortic lymphadenectomy
  Groups: Group with lymphadenectomy

SUMMARY:
The purposes of this study are

* to determine the prevalence, size and impact on quality of life of lymphedema of the lower extremities after primary radical surgery with hysterectomy +/- pelvic - and paraaortic lymphadenectomy in women with endometrial uterine carcinoma FIGO (International Federation of Gynecology and Obstetrics) stage 1 and 2
* to analyze risk factors for development of lymphedema in this specific group of patients.

Our hypotheses are that women who have lymphadenectomy more often suffer from lymphedema, subjectively and objectively, and have an impaired quality of life.

This is a Swedish multicenter study carried out in 17 departments of Obstetrics and Gynecology and in 3 departments of Oncology. All participants are treated according to the Swedish National Guidelines for Endometrial Cancer.

130 women with endometrial cancer who have a hysterectomy with lymphadenectomy (high-risk endometrial carcinomas) and 130 women with endometrial cancer who have a hysterectomy without lymphadenectomy (low-risk endometrial carcinomas) are prospectively enrolled in the study.

The participants are examined preoperatively and on 3 occasions postoperatively, i.e. 4-6 weeks , 6 months and 12 months postoperatively.

Determination of occurrence of lymphedema of the lower extremities are determined objectively by 1) a standardized clinical evaluation according to Bruna et al.[1] and 2) determining the leg volume according to the cone model by Sitzia [2] by systematically measuring of leg circumferences. In addition, occurrence of lymphedema is measured subjectively by the participants.

On the same four occasions as the leg circumference measurements are conducted the patients complete two generic health related quality of life forms (the EuroQol EQ-5D and the Short-Form 36 SF-36) and the condition specific quality of life form for limb lymphedema (LYMQOL).

Demographic and clinical data are systematically collected until one year postoperatively including occurrence of complications and given adjuvant oncological therapy such as chemo- and radiation therapy.

On each occasion of clinical control a vaginal ultrasound examination is carried out in order to register pelvic and abdominal lymphocele formation or lymphatic fluid effusion intraabdominally.

DETAILED DESCRIPTION:
Not included

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Women with endometrial carcinoma preoperatively evaluated to be uterine cancer FIGO stage1 or 2 who are planned for primary radical surgery including simple or radical hysterectomy, bilateral salpingoophorectomy,+/- pelvic and paraaortic lymphadenectomy and +/- omentectomy with curative intention.
* WHO performance status ≤ 2.
* Understand and speak Swedish fluently
* Accept to participate in the study by giving verbal and written informed consent.

Exclusion Criteria:

* Sarcoma of the uterus
* Previous pelvic or paraaortic lymphadenectomy.
* Previous having had pelvic radiation therapy.
* Ongoing treatment of arterial or venous insufficiency of the lower limbs
* Congenital or acquired malformations in the lymphatic system.
* Ongoing or previous treatment of lymphedema of the upper or lower limbs.
* Physically disability which impair mobilisation immediately postoperatively.
* Severe psychiatric disease and untreated mild/moderate psychiatric disease.
* Mentally retarded to a degree so she does not understand the meaning of the participation or cannot fill in the questionnaires.or the physician finds it ethically doubtful to enroll the patient in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women admitted to the participating clinics for primary surgery of endometrial carcinoma FIGO stage 1 and 2 will be asked to participate in the study.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Change in leg volume from baseline (preoperatively) to 4-6 weeks postoperatively | 4-6 weeks after the primary surgery
  Leg volume is determined by the cone model according to Sitzia by measuring leg circumferences systematically.
Change in leg volume from baseline (preoperatively) to 6 months postoperatively | 6 months after the primary surgery
  Leg volume is determined by the cone model according to Sitzia by measuring leg circumferences systematically.
Change in leg volume from baseline (preoperatively) to 12 months postoperatively | 12 months after the primary surgery
  Leg volume is determined by the cone model according to Sitzia by measuring leg circumferences systematically.

SECONDARY OUTCOMES:
Change in quality of life assessment from baseline (preoperatively) to 4-6 weeks postoperatively | 4-6 weeks from the primary surgery
  Quality of life measured by means of The EuroQol (EQ-5D), the Short-Form 36 (SF-36) and the condition specific quality of life form LYMQOL.
Change in quality of life assessment from baseline (preoperatively) to 6 months postoperatively | 6 months from the primary surgery
  Quality of life measured by means of The EuroQol (EQ-5D), the Short-Form 36 (SF-36) and the condition specific quality of life form LYMQOL.
Change in quality of life assessment from baseline (preoperatively) to 12 months postoperatively | 12 months from the primary surgery
  Quality of life measured by means of The EuroQol (EQ-5D), the Short-Form 36 (SF-36) and the condition specific quality of life form LYMQOL.
Percentage of participants with an increase in leg volume of > 15% 12 months postoperatively | 12 months after the primary surgery
Percentage of participants who states they have lymphedema | 12 months from the primary surgery
  Occurrence of lymphedema subjectively graded as 2 or more on an ordinal scale from 1 to 4. 1 express no swelling of the legs and 4 express severe swelling.

OTHER OUTCOMES:
Risk factors for lymphedema after primary surgery with lymphadenectomy for endometrial cancer | Within 12 months after the surgery
  Risk factors defined in terms of number of lymphnodes removed, site of lymphnodes, peri- and postoperative complications, adjuvant chemotherapy, adjuvant radiation therapy, age, histopathological subtype, surgical FIGO stage, DNA-ploidy status of the tumor, comorbidity and relapse of the cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjölhede, MD, PhD, Study Chair — Dept of Obs/Gyn, University Hospital, Linköping; Per Rosenberg, MD,PhD, Study Chair — Dept of Oncology, University Hospital, Linköping; Gabriel Lindahl, MD, Study Chair — Dept of Oncology, University Hospital, Linköping; Eva Ahlner, RPT, Study Chair — Dept of Oncology, University Hospital, Linköping; Janusz Marcickiewicz, MD, PhD, Study Chair — Dept of Obs/Gyn, Region Halland Varberg Hospital, Varberg; Karin Stålberg, MD, PhD, Study Chair — Dept of Obs/Gyn, Univeristy Hospital, Uppsala; Ulrika Ottander, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Norrlands University Hospital, Umeå; Kristina Aglund, MD, PhD, Principal Investigator — Dept of Oncology, Norrlands University Hospital, Umeå; Åsa Åkesson, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Sahlgrenska University Hospital, Göteborg; Eva Blank, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Norra Älvsborg County Hospital in Trollhättan, Trollhättan; Lars Högström, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Södra Älvsborgs Hospital, Borås; Eva Rundqvist, MD, Principal Investigator — Dept of Obs/Gyn, Blekinge Hospital, Karlskrona; Margareta Lood, MD, Principal Investigator — Dept of Obs/Gyn, Central Hospital, Karlstad; Lotta Andreen, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Central Hospital, Sundsvall; Peter Smith, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Central Hospital, Gävle; Åsa Nyberg, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Central Hospital, Falun; Lisbeth Liest, MD, Principal Investigator — Dept of Obs/Gyn, Highland Hospital, Eksjö; Gunnel Lindell, MD, PhD, Principal Investigator — Dept of Obs/Gyn, Kalmar County Hospital, Kalmar; Anders Rosenmüller, MD, Principal Investigator — Dept of Obs/Gyn, Västervik County Hospital, Västervik
Locations (16):
- Sweden (16):
  - Highland hospital, Eksjö, Jonkopings Län
  - Falu Central Hospital, Falun
  - Gävle County Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Region Halland Halmstad Hospital, Halmstad
  - County Hospital in Kalmar, Kalmar
  - Blekinge Hospital, Karlskrona
  - Karlstad Central Hospital, Karlstad
  - Linkoping University Hospital, Linköping
  - Södra Älvborgs Sjukhus, Skövde
  - Sundsvall Hospital, Sundsvall
  - Norra Älvborgs Hospital, Trollhättan
  - Norrlands University Hospital, Umeå
  - Akademiska University Hospital, Uppsala
  - Region Halland Varberg hospital, Varberg
  - Västervik County Hospital, Västervik

REFERENCES:
- [Background] Miller AJ, Bruna J, Beninson J. A universally applicable clinical classification of lymphedema. Angiology. 1999 Mar;50(3):189-92. doi: 10.1177/000331979905000302. PMID 10088797
- [Background] Sitzia J. Volume measurement in lymphoedema treatment: examination of formulae. Eur J Cancer Care (Engl). 1995 Mar;4(1):11-6. doi: 10.1111/j.1365-2354.1995.tb00047.x. PMID 7620649